CLINICAL TRIAL: NCT05901649
Title: Prospective, Multi-Country, Observational Study of Clinical Outcomes for Participants With Metastatic Hormone Sensitive Prostate Cancer (mHSPC) Treated With ADT Plus Apalutamide or Enzalutamide Under Routine Clinical Practice (ArtemisPRO)
Brief Title: A Study for the Participants With Metastatic Hormone Sensitive Prostate Cancer (mHSPC) Treated With Androgen Deprivation Therapy (ADT) Plus Apalutamide or Enzalutamide
Acronym: ArtemisPRO
Status: Active, not recruiting | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109320; 56021927PCR4031 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer
MeSH Terms: interventions — apalutamide; enzalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Apalutamide Plus Androgen Deprivation Therapy (ADT): Participants with metastatic hormone-sensitive prostate cancer (mHSPC) will be observed who are being treated with apalutamide under clinical practice setting. Only data available per routine clinical practice will be collected within this study.
  Interventions: Drug: Apalutamide
- Enzalutamide Plus Androgen Deprivation Therapy (ADT): Participants with metastatic hormone-sensitive prostate cancer (mHSPC) will be observed who are being treated with enzalutamide under clinical practice setting. Only data available per routine clinical practice will be collected within this study.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Apalutamide — No interventions will be administered as a part of this study. Participants will receive apalutamide as per their routine clinical practice.
  Other Names: ERLEADA
  Groups: Apalutamide Plus Androgen Deprivation Therapy (ADT)
Drug: Enzalutamide — No interventions will be administered as a part of this study. Participants will receive enzalutamide as per their routine clinical practice.
  Other Names: XTANDI
  Groups: Enzalutamide Plus Androgen Deprivation Therapy (ADT)

SUMMARY:
The purpose of this study is to assess the real-world outcomes differences between apalutamide or enzalutamide plus androgen deprivation therapy (ADT) for the treatment of participants with metastatic hormone-sensitive prostate cancer (mHSPC).

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically or cytologically-confirmed diagnosis of adenocarcinoma of the prostate
* Must have documented metastatic hormone-sensitive prostate cancer (mHSPC)
* Must have agreed with the treating physician the initiation of either apalutamide or enzalutamide (plus androgen deprivation therapy [ADT]) treatment, per the treating physician's decision, prior to enrollment into the study
* Must sign, and/or their legally acceptable representative where applicable must sign, a participation agreement/ informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements
* Must have baseline prostate-specific antigen (PSA) captured within 30 days prior to the first administration of apalutamide or enzalutamide
* Must agree to complete patient-reported outcomes (PROs) during the study, including the baseline ones collected before the first administration of apalutamide or enzalutamide

Exclusion Criteria:

* Has already received or is currently receiving either apalutamide or enzalutamide, or any other novel hormonal treatments (including but not limited to abiraterone acetate and darolutamide)
* Is currently receiving an active treatment for prostate cancer as part of an interventional study
* Has a progression under ADT treatment (and thus became castrate-resistant) prior to start of apalutamide or enzalutamide treatment
* Has received ADT treatment for mHSPC for more than 2 months prior to apalutamide or enzalutamide treatment initiation or ADT treatment was administered for earlier disease stages within the last 12 months prior to apalutamide or enzalutamide treatment initiation
* Has received prior docetaxel for the treatment of mHSPC
* Participants is not treated in line with current Summary of Product Characteristics for apalutamide or enzalutamide

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with high-risk metastatic hormone-sensitive prostate cancer (mHSPC) who will be treated with either apalutamide or enzalutamide plus androgen deprivation therapy (ADT) under routine clinical practice will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Prostate-specific Antigen (PSA) Level <0.2 ng/mL at Month 3 | At month 3
  Percentage of participants with PSA level less than (<)0.2 nanogram per milliliter (ng/mL) at month 3 will be reported.
Health-Related Quality of Life (HRQoL) as Assessed by Partial European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Questionnaire | Up to 30 Months
  HRQoL of the participants will be assessed as partial EORTC QLQ-C30 questionnaire. EORTC QLQ-C30 scale scores range from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptom.
Cognitive Functioning as Assessed by Partial Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) Questionnaire | Up to 30 Months
  Cognitive function of the participants will be measured by the partial FACT-Cog (Version 3) questionnaire. The FACT-Cog score ranges from scale 0-148. The higher the total score, the better the cognitive function.
Fatigue as Assessed by Brief Fatigue Inventory-Short Form (BFI-SF) Questionnaire | Up to 30 Months
  Participant fatigue will be assessed by the BFI-SF questionnaire. The BFI-SF score range from scale 0-10. Scores are categorized as Mild (1-3), Moderate (4-6), and Severe (7-10).
Prostate-specific Antigen (PSA) Anxiety as Assessed by Memorial Anxiety Scale for Prostate Cancer (MAX-PC) Questionnaire | Up to 30 Months
  PSA anxiety of the participant will be assessed by the MAX-PC questionnaire. The MAX-PC total score ranges from scale 0 to 54. The MAX-PC is divided into three subscales: a) prostate cancer anxiety (PCA) range from 0 to 33, b) Prostate-Specific Antigen Anxiety (PSAA) ranges from 0 to 9, and c) fear of recurrence (FOR) ranges from 0 to 12.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (53):
- Austria (2):
  - Akh Wien, Vienna
  - Klinikum Wels Grieskirchen, Wels
- France (16):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Acquitaine, Bordeaux
  - Clinique Pasteur- Lanroze, Brest
  - Hopital Michallon CHU Grenoble Alpes, La Tronche
  - Hôpital Edouard Herriot, Lyon
  - Centre d'oncologie de Gentilly, Nancy
  - CHU Nimes, Nîmes
  - Hopital Europeen Georges-Pompidou, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Rene Dubos Pontoise, Pontoise
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Centre Hospitalier Prive, Saint-Grégoire
  - Clinique Sainte Anne, Strasbourg
  - Hopital Foch, Suresnes
  - CHU de Toulouse, Toulouse
- Germany (8):
  - Urologie Dierdorf, Dierdorf
  - St. Elisabeth Hospital Leipzig, Dresden
  - Urologicum Duisburg, Duisburg
  - Urologisches Zentrum Mittelhessen, Gladenbach
  - Praxis Dr. Serkan Filiz, Hamburg
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
- Greece (7):
  - Alexandra General Hospital of Athens, Athens
  - Anticancer Oncology Hospital of Athens Agios Savvas, Athens
  - Attikon University General Hospital of Attica, Athens
  - General Oncology Hospital of Kifisias "Agioi Anargyroi, Athens
  - University Hospital of Heraklion, Heraklion
  - University General Hospital of Rio Patras, Pátrai
  - Papageorgiou General Hospital Of Thessaloniki, Thessaloniki
- Spain (9):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Torrecardenas, Almería
  - Hosp. Puerta Del Mar, Cadiz
  - Hosp. Gral. Univ. de Castellon, Castellon
  - Hosp. Univ. Lucus Augusti, Lugo
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Univ. de Canarias, San Cristóbal de La Laguna
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Univ. I Politecni La Fe, Valencia
- United Kingdom (11):
  - Frimley Health NHS Foundation Trust, Berkshire
  - Royal Cornwall Hospitals NHS Trust - Royal Cornwall Hospital, Cornwall
  - Torbay Hospital-Devon, Devon
  - Dorset County Hospital Nhs Foundation Trust, Dorchester
  - Royal Surrey County Hospital NHS Trust, Guildford
  - University College London Hospitals Nhs Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Pennine Care Nhs Foundation Trust, Oldham
  - Scunthorpe General Hospital, Scunthorpe
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - University Hospitals Sussex NHS Foundation Trust Worthing Hospital, Worthing

IPD SHARING:
Plan to Share IPD: No